CLINICAL TRIAL: NCT02401386
Title: A Randomized Controlled Trial of Eight Brocades (Ba Duan Jin) to Improve Quality of Life in Patients With Fibromyalgia
Brief Title: Eight Brocades (Ba Duan Jin) for Treating Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Juan Jiao, Associate chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z141107002514094
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Eight Brocades; Baduanjin; Qigong; Pain severity
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EB group (Experimental): Trained and guided by EB certified physicians, patients in EB group received closely supervised, group-format EB program and practiced EB for one hour, twice weekly for 12 weeks in the Guang'anmen Hospital.
  Interventions: Behavioral: The Eight Brocades
- Control group (No Intervention): The participants in usual therapy-controlled group will stay on their previous treatment through 12 weeks. As compensation, they will be invited to receive LEB training for 12 weeks after the end of the study.

INTERVENTIONS:
Behavioral: The Eight Brocades — Patients received closely supervised, group-format EB program and practiced EB revised by Chinese Medicine Master Zhi-zheng Lu for one hour, twice weekly for 12 weeksmovements, a review of principles, and breathing techniques in EB. Participants will be asked to practice EB at home for at least 16 minutes each day which is how long it takes to complete an EB exercise, using an instructional Digital Video Disc. The program will be taught by experienced EB masters.
  Arms: EB group

SUMMARY:
In this randomized, usual therapy-controlled study, 62 patients with fibromyalgi (FM) were recruited with a ratio of 1:1. Trained and guided by Eight Brocades (EB) certified physicians, participant practiced EB one hour, twice a week for 12 weeks. Evaluation will be based on standard scales of pain, FM symptoms severity, degree of fatigue, depression, sleep quality and quality of life.

DETAILED DESCRIPTION:
The EB, also written as Ba Duan Jin, or Baduanjin, or Eight-Section Brocade, is a set of Qigong exercises that originated in China and date back thousands of years. It is a mind-body practice that combines meditation with slow, gentle, graceful movements, as well as deep breathing and relaxation, to move vital energy (or qi) throughout the body and is practiced as a rehabilitation exercise for various kinds of diseases. It is considered a complex, multicomponent intervention that integrates physical, psychosocial, emotional, spiritual, and behavioral elements. Participants in the EB group received a modified EB adapted by Chinese Medicine Master Zhi-zheng Lu, which was added several joint exercise movements to the traditional EB forms to specifically tailor it for patients with rheumatic diseases.

FM is a common and complex clinical syndrome characterized by chronic and widespread musculoskeletal pain, fatigue, sleep disturbance, and physical and psychological impairment. Evidence-based guidelines suggest that exercise is beneficial for FM and has been advocated as a core component of its treatment. Because of EB's mind-body attributes and it is easy to learn, we assume that it could be well suited for the treatment of FM.

Patients enrolled in this trial will be randomly allocated into one of two groups: EB group and usual therapy-controlled group. Patients will be evaluated at baseline, at week 4, 8 and 12. The primary outcome measure was a Visual Analogue Scales for pain (PVAS). Secondary outcome measures included the following: the Revised FM Impact Questionnaire (FIQR), the Multidimensional Assessment of Fatigue (MAF), the Pittsburgh Sleep Quality Index (PSQI), the Beck Depression Inventory (BDI), the Perceived Stress Scale (PSS), and the Tender Points Count (TPC).

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 years or older.

  * Fulfills the American College of Rheumatology (ACR) 1990 classification criteria for FM.
  * On a stable variety and dosage of pharmacologic for FM ≥4 weeks

Exclusion Criteria:

* • Prior experience with EB or other similar types of Complementary and Alternative Medicine in the past 1 year such as Qi gong, Tai Chi and yoga since these share some of the principles of EB.

  * Dementia, cancer, or other serious medical conditions limiting ability to participate in the Eight Brocades or strength training, as determined by the study physicians.
  * Any other diagnosed medical condition known to contribute to FM symptomatology that is not under adequate control for the study period such as thyroid disease, inflammatory arthritis, systemic lupus erythematosus, rheumatoid arthritis, myositis, vasculitis or Sjogren's syndrome.
  * Positive urine pregnancy test at baseline or planning pregnancy within the study period.
  * Reside >70 miles from the research site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The change of Visual Analogue Scales for pain (PVAS) from baseline to 12 weeks. | baseline, 4 weeks, 8 weeks, 12 weeks
The change of Fibromyalgia Impact Questionnaire (FIQ) from baseline to 12 weeks | baseline, 4 weeks, 8 weeks, 12 weeks

SECONDARY OUTCOMES:
The change of the Short Form-36 Health Status Questionnaire (SF-36) from baseline to 12 weeks | baseline, 4 weeks, 8 weeks, 12 weeks
The change of Multidimensional Assessment Fatigue (MAF) from baseline to 12 weeks | baseline, 4 weeks, 8 weeks, 12 weeks
The change of Beck depression inventory (BDI) from baseline to 12 weeks | baseline, 4 weeks, 8 weeks, 12 weeks
The change of Perceived Stress Scale (PSS) from baseline to 12 weeks | baseline, 4 weeks, 8 weeks, 12 weeks
The change of Pittsburgh sleep quality index (PSQI) from baseline to 12 weeks | baseline, 4 weeks, 8 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juan Jiao, M.D.,PhD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China